CLINICAL TRIAL: NCT02650336
Title: Aging Biomakers and ConTrast Induced Nephropathy (ACTIN) Trial
Acronym: ACTIN
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiao-dong Zhuang, department of cardiology, first affiliated hoapital of SYSU, Sun Yat-sen University
Other Study IDs: ACTIN-sysu
Record Dates: First submitted 2016-01-03; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Contrast Induced Nephropathy
MeSH Terms: interventions — Contrast Media

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Morning blood samples were received from all volunteers after an 8-h overnight fast. The investigators obtained the blood samples used to measure preoperative serum uric acid, baseline serum creatinine (SCr) (prior to the pre-procedural hydration), blood urea nitrogen (BUN), fasting blood glucose, random blood glucose, electrolytes before PCI, serum lipids, albumin, hemoglobin, and other standard clinical parameters. Blood samples were left to clot for one hour and then centrifuged at 1500 ×g for 10 min. Plasma samples were accumulated and stored at -80 °C until analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CIN proup: The occurrence of CIN was defined as an increase in serum creatinine of 0.5 mg/dL above the baseline value within 48-72 h after PCI. Follow-up SCr and BUN levels were measured 1, 2, and 3 days after the procedure.
  Interventions: Drug: contrast
- control group: The occurrence of CIN was defined as an increase in serum creatinine of 0.5 mg/dL above the baseline value within 48-72 h after PCI. Follow-up SCr and BUN levels were measured 1, 2, and 3 days after the procedure.
  Interventions: Drug: contrast

INTERVENTIONS:
Drug: contrast — a substance used to enhance the contrast of structures or fluids within the body in medical imaging. It is commonly used to enhance the visibility of blood vessels and the gastrointestinal tract
  Other Names: low-osmolar, non-ionic contrast medium

SUMMARY:
Biomarkers such as kidney injury molecule-1 (KIM-1) and neutrophil gelatinase-associated lipocalin (NGAL) have been used for the early diagnosis of AKI, although with no definitive results. The investigators explored the association between plasma aging biomakers such as sklotho and contrast induced nephropathy in patients undergoing percutaneous coronary intervention (PCI) with contrast injection.

DETAILED DESCRIPTION:
Acute kidney injury represents an important clinical problem in hospitalized patients, with persistently high rates of mortality and morbidity. With an ever-increasing number of patients receiving intravascular injection of iodinated contrast media worldwide, contrast induced nephropathy (CIN) has become the third leading cause of hospital-acquired AKI. Approximately half of these cases are in patients undergoing cardiac catheterization procedures.

The prevention and early intervention of CIN has been hampered mainly by the lack of a consensus definition and the paucity of early predictive biomarkers to accurately identify high-risk patients. CIN is most frequently defined as an increase in serum creatinine (sCr) by 25-50% above the baseline, generally occurring within the first 24 h after contrast exposure, in the absence of other causes. However, sCr is an unreliable indicator during acute changes in kidney function, and alterations in sCr levels are not particularly sensitive or specific for small changes in the glomerular filtration rate (GFR)e, gender, race and intravascular volume. Biomarkers such as kidney injury molecule-1 (KIM-1) and neutrophil gelatinase-associated lipocalin (NGAL) have been used for the early diagnosis of AKI, although with no definitive results.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older undergoing planed PCI were prospectively recruited

Exclusion Criteria:

* Pregnancy
* Lactation
* Sepsis
* The intravascular administration of a contrast medium within the past 7 days, nephroprotective drug treatment (e.g., N-acetylcysteine, theophylline, sodium bicarbonate, prostaglandin E1)
* Nephrotoxic drug intake (e.g., non-steroidal anti-inflammatory drugs, metformin, aminoglycosides, cisplatin) within the past 7 days
* A history of serious allergic to contrast media
* Renal transplantation
* End-stage renal disease necessitating dialysis
* Severe concomitant disease of other systems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older undergoing planed PCI at the institution of first affiliated hospital of SYSU were prospectively recruited between May 2014 and July 2015. The exclusion criteria were pregnancy, lactation, sepsis, the intravascular administration of a contrast medium within the past 7 days, nephroprotective drug treatment (e.g., N-acetylcysteine, theophylline, sodium bicarbonate, prostaglandin E1), nephrotoxic drug intake (e.g., non-steroidal anti-inflammatory drugs, metformin, aminoglycosides, cisplatin) within the past 7 days, a history of serious allergic to contrast media, renal transplantation, end-stage renal disease necessitating dialysis, and severe concomitant disease of other systems.
Sampling Method: Non-Probability Sample
Enrollment: 592 (Actual)
Dates: Start 2013-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The association between plasma aging biomakers and contrast induced nephropathy | 48-72 hours
  The plasma concentrations human soluble a-Klotho levels were measured by Enzyme Linked Immunosorbent Assay (ELISA) (Immuno-Biologic Laboratories Co., Ltd. Japan). This novel method detects sklotho using a monoclonal antibody with high affinity to the human a-Klotho protein.Hs-CRP was tested with a Beckman Coulter Immage immunobiochemistry system (USA) using nephelometry (unit: mg/L). Creatinine clearance (CrCl) was calculated by applying the Cockcroft- Gault formula to the serum creatinine concentration.

SECONDARY OUTCOMES:
The association between plasma aging biomakers and in-hospital MACE in patients undergoing percutaneous coronary intervention (PCI) with contrast injection. | 30 days, 1 year
  In-hospital major adverse cardiovascular events (MACE):defined as (1) death, (2) nonfatal myocardial infarction, or (3) target vessel revascularization. Myocardial infarction was diagnosed by a rise in the creatine kinase level to more than twice the upper normal limit with an increased creatine kinase-MB. Target lesion revascularization was defined as a repeat intervention (surgical or percutaneous) to treat a luminal stenosis within the stent or in the 5-mm distal or proximal segments adjacent to the stent. Target vessel revascularization was defined as a reintervention driven by any lesion located in the same epicardial vessel. Thrombotic stent occlusion was angiographically documented as a complete occlusion (TIMI flow 0 or 1) or a flow-limiting thrombus (TIMI flow 1 or 2) of a previously successfully treated artery.

CONTACTS AND LOCATIONS:
Overall Officials: zhimin du, MD, Principal Investigator — fitst affiliated hospital of SYSU
Locations (1):
- Xiaodong Zhaung, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No